CLINICAL TRIAL: NCT04554043
Title: A Randomized, Double-blind, Dose-escalation, Placebo-controlled Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Oral Doses of SHR7280 Tablets in Healthy Subjects.
Brief Title: The PK/PD Study of SHR7280 Tablets in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR7280-103
Record Dates: First submitted 2020-08-31; First posted 2020-09-18 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- SHR7280 dose 1(male) (Experimental): oral administration for 14 days,Phase I(PART 1)
  Interventions: Drug: SHR7280; Drug: Placebo oral tablet
- SHR7280 dose 2(male) (Experimental): oral administration for 14 days,Phase I(PART 1)
  Interventions: Drug: SHR7280; Drug: Placebo oral tablet
- SHR7280 dose 3(male) (Experimental): oral administration for 14 days,Phase I(PART 1)
  Interventions: Drug: SHR7280; Drug: Placebo oral tablet
- SHR7280 dose 4(male) (Experimental): oral administration for 14 days,Phase I(PART 1)
  Interventions: Drug: SHR7280; Drug: Placebo oral tablet
- SHR7280 dose 5(male) (Experimental): oral administration for 14 days,Phase I(PART 1)
  Interventions: Drug: SHR7280; Drug: Placebo oral tablet
- SHR7280 dose 1(female) (Experimental): oral administration for 21 days,Phase I(PART 2)
  Interventions: Drug: SHR7280; Drug: Placebo oral tablet
- SHR7280 dose 2(female) (Experimental): oral administration for 21 days,Phase I(PART 2)
  Interventions: Drug: SHR7280; Drug: Placebo oral tablet
- SHR7280 dose 3(female) (Experimental): oral administration for 21 days,Phase I(PART 2)
  Interventions: Drug: SHR7280; Drug: Placebo oral tablet
- SHR7280 dose 4(female) (Experimental): oral administration for 21 days,Phase I(PART 2)
  Interventions: Drug: SHR7280; Drug: Placebo oral tablet
- SHR7280 dose 6(male) (Experimental): oral administration for 14 days,Phase I(PART 1)
  Interventions: Drug: SHR7280; Drug: Placebo oral tablet
- SHR7280 dose 7(male) (Experimental): oral administration for 14 days,Phase I(PART 1)
  Interventions: Drug: SHR7280; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: SHR7280 — treatment
Drug: Placebo oral tablet — blank control

SUMMARY:
The primary objective of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of SHR7280 tablets in healthy subjects.

DETAILED DESCRIPTION:
GNRH antagonists can be used to treat sex hormone-dependent diseases, and SHR7280 is an oral GNRH antagonist. The purpose of this study is to observe the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple oral doses of SHR7280 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

PART 1:

1. Healthy males , aged 18-65;
2. BMI 18 ~ 30 kg/m2;
3. Subjects in general good health. No clinically significant findings in Physical examination and auxiliary examination.

PART 2:

1. premenopausal females, aged 18-45;
2. BMI 18 ~ 30 kg/m2;
3. Subjects in general good health. No clinically significant findings in Physical examination and auxiliary examination.

Exclusion Criteria:

PART 1

1. Testosterone (T) < 12 nmol/L;
2. ALT or AST or total bilirubin exceeds the upper limit of normal;
3. Those with positive nicotine test and alcohol breath test before administration, and those with positive drug screening before administration;
4. Use of any medication within 1 month before administration; or use of medication that does not exceed 5 half-lives, whichever is longer;
5. Subjects with chronic diseases or serious diseases that affect drug absorption, distribution, metabolism and excretion;
6. Blood donation or donation of blood components within 1 month before screening, or loss of blood equivalent to at least 200 mL, or transfusion within 2 months;
7. Use of GnRH agonists and GnRH antagonists within 6 months before screening and use of any androgens and antiandrogens within 5 half-lives before screening;
8. Subjects with severe infection, severe trauma or major surgery within 6 months before screening;
9. Positive results of infectious disease screening .
10. Allergic constitution or allergy to two or more kinds of food and drugs, including known history of allergy to the study drug or any component of the study drug.

PART 2:

1. Pregnant or breast feeding;
2. FSH≥25U/L;
3. Positive serum pregnancy test (serum β-HCG test) result;
4. Abnormal uterine bleeding within 3 months prior to screening
5. ALT or AST or total bilirubin exceeds the upper limit of normal;
6. Those with positive nicotine test and alcohol breath test before administration, and those with positive drug screening before administration;
7. Use of any medication within 1 month before administration; or use of medication that does not exceed 5 half-lives, whichever is longer;
8. Subjects with chronic diseases or serious diseases that affect drug absorption, distribution, metabolism and excretion;
9. Blood donation or donation of blood components within 1 month before screening, or loss of blood equivalent to at least 200 mL, or transfusion within 2 months;
10. GnRH agonist use 6 months prior to Screening and GnRH antagonist or any sex hormone use 2 months prior to Screening.
11. Subjects with severe infection, severe trauma or major surgery within 6 months before screening
12. Positive results of infectious disease screening .
13. Allergic constitution or allergy to two or more kinds of food and drugs, including known history of allergy to the study drug or any component of the study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse events | Pre-dose to 28±2 days after dose administration
  Part 1 and Part 2

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUCτ) after the first dose of SHR7280; | At pre-defined intervals from initial dose through final study visit( 28±2 days after dose administration)
  Part 1 and Part 2
Maximum observed serum concentration (Cmax) after the first dose of SHR7280; | At pre-defined intervals from initial dose through final study visit (28±2 days after dose administration)
  Part 1 and Part 2
Time to maximum observed serum concentration (Tmax) after the first dose of SHR7280; | At pre-defined intervals from initial dose through final study visit (28±2 days after dose administration)
  Part 1 and Part 2
Time to elimination half-life (T1/2) ; | At pre-defined intervals from initial dose through final study visit (28±2 days after dose administration)
  Part 1 and Part 2
Apparent total clearance(CL/F) of the drug from plasma after last morning dose of SHR7280; | At pre-defined intervals from initial dose through final study visit (28±2 days after dose administration)
  Part 1 and Part 2
Apparent volume of distribution(Vz/F) after last morning dose of SHR7280; | At pre-defined intervals from initial dose through final study visit (28±2 days after dose administration)
  Part 1 and Part 2
Maximum observed serum concentration (Cmax) after last morning dose of SHR7280; | At pre-defined intervals from initial dose through final study visit (28±2 days after dose administration)
  Part 1 and Part 2
Time to maximum observed serum concentration (Tmax) after last morning dose of SHR7280; | At pre-defined intervals from initial dose through final study visit (28±2 days after dose administration)
  Part 1 and Part 2
Trough observed serum concentration (Ctrough) after last morning dose of SHR7280; | At pre-defined intervals from initial dose through final study visit (28±2 days after dose administration)
  Part 1 and Part 2
Accumulation Factor（Racc）after last morning dose of SHR7280; | At pre-defined intervals from initial dose through final study visit (28±2 days after dose administration)
  Part 1 and Part 2
Area under the plasma concentration versus time curve (AUCτ) after last morning dose of SHR7280; | At pre-defined intervals from initial dose through final study visit (28±2 days after dose administration)
  Part 1 and Part 2
Endocrine Parameters: Testosterone | At pre-defined intervals from initial dose through final study visit (28±2 days after dose administration)
  Part 1
Endocrine Parameters: Estuarial | At pre-defined intervals from initial dose through final study visit (28±2 days after dose administration)
  Part 2
Endocrine Parameters:Progesterone | At pre-defined intervals from initial dose through final study visit (28±2 days after dose administration)
  Part 2
Endocrine Parameters: Luteinizing hormone | At pre-defined intervals from initial dose through final study visit (28±2 days after dose administration)
  Part 2
Endocrine Parameters: Follicle stimulating hormone | At pre-defined intervals from initial dose through final study visit (28±2 days after dose administration)
  Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, PhD, Principal Investigator — Hospital of Qingdao University
Locations (1):
- Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
Hengrui shall own the exclusive rights to all results, data, findings, radiological & diagnostic images, discoveries, inventions & specifications, whether patentable or not, that are originated, conceived, derived, produced, discovered, invented or otherwise made by Center, PI and/or Study Team Physicians and/or Members in connection with the performance of the Study (i.e. Results).

REFERENCES:
- [Derived] Li X, Sun F, Zhang X, Lin P, Shen K, Shen Y, Ma L, Cao Y, Wang C. Safety, pharmacokinetics, and pharmacodynamics of SHR7280, an oral gonadotropin-releasing hormone receptor antagonist, in healthy men: a randomized, double-blind, placebo-controlled phase 1 study. BMC Med. 2023 Apr 3;21(1):129. doi: 10.1186/s12916-023-02834-6. PMID 37013610
- [Derived] Xu Y, Hu W, Li J, Jiang X, Shi P, Shen K, Shen Y, Ma L, Cao Y. Safety, pharmacokinetics, and pharmacodynamics of SHR7280, an oral gonadotropin-releasing hormone antagonist in healthy premenopausal women. Front Pharmacol. 2022 Nov 23;13:1027648. doi: 10.3389/fphar.2022.1027648. eCollection 2022. PMID 36506562